CLINICAL TRIAL: NCT02007902
Title: Early Plasma Protein Levels and Neonatal Hemodynamics: a Prospective Evaluation in Very Preterm Infants
Brief Title: Plasma Protein Levels and Very Preterm Birth
Acronym: ProHémie
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: INSERM CIE1, Dijon, 21000, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2013/CHU/02; 2013-A00090-45 (Other: Agence Nationale de Sécurité du Médicament)
Record Dates: First submitted 2013-11-25; First posted 2013-12-11 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Very Preterm Infants
Keywords: Preterm baby; Total plasma protein; Albumin; Hemodynamic disturbances; Perfusion; Near Infra Red Spectroscopy (NIRS); Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Very preterm babies: Observational model: cohort
  Interventions: Other: Evaluation of the relationship plasma protein levels - neonatal hemodynamics

INTERVENTIONS:
Other: Evaluation of the relationship plasma protein levels - neonatal hemodynamics — * Patient inclusion at birth
  * Total plasma protein values measurement on cord blood sample at birth
  * Hemodynamic evaluation at 6 hours after birth with colour doppler echocardiography and organ blood flow colour doppler
  * Total plasma protein and albumin values measurement on plasma sample at 12 hours after birth
  * Blood pressure, heart rate, O2 saturation, capillary refill time, rSO2 [regional (cerebral and somatic) tissue oxygenation by NIRS - near infrared spectroscopy] will be monitored over 24 hours after birth.

SUMMARY:
The primary aim of this study is to investigate the relationship between early plasma protein levels and hemodynamics in very preterm infants during postnatal transition. Secondary aims are the following: i) to evaluate maternal and neonatal factors affecting plasma protein level at birth; ii) to evaluate the relationship between plasma protein level and albumin level on the first day of life; iii) to evaluate the association between early hypoproteinemia and neonatal mortality and morbidity in very preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Parents written informed consent
* Birth at less than 32 weeks of gestational age
* Birth in a III level delivery facility at Reunion Island

Exclusion Criteria:

* Major congenital abnormalities

Ages: 1 Minute to 1 Hour | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Very preterm infants with birth at less than 32 weeks of gestational age
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Evidence of clinical hemodynamic disturbances defined by arterial hypotension (non-invasive measure of MAP - mmHg - pathological for gestational age) or measured at organ colour doppler, echocardiography or NIRS | about 6 hours after birth

SECONDARY OUTCOMES:
plasma protein | at 1 second after birth (cord blood sample)
  plasma protein level on cord blood sample depending on maternal and neonatal variables
Albumin level | At 12 hours after birth
Mortality rate | patients will be followed for the duration of hospital stay, that is an average of 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Iacobelli, Principal Investigator — CHU de La Réunion -Site du GHSR; Sylvain Samperiz, MD, Principal Investigator — CHU de La Réunion - Hôpital Félix Guyon
Locations (2):
- France (2):
  - Centre Hopsitalier Universitaire de La Réunion, Saint-Denis, La Réunion
  - Centre Hospitalier de La Réunion, Saint-Pierre, La Réunion